CLINICAL TRIAL: NCT04480294
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics, Pharmacodynamics of Oral HRS5091 in Healthy Subjects With Single or Multiple Dose and Chronic Hepatitis B Patients With Multiple Dose, and Food Effects of HRS5091 in Healthy Subjects
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Oral HRS5091 in Healthy Subjects and Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HRS5091-101
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part 1a Treatment group 1 (Experimental): Intervention: Drug1: HRS5091, dose 1; Drug2: Placebo Healthy subjects
  Interventions: Drug: HRS5091
- Part 1a Treatment group 2 (Experimental): Intervention: Drug1: HRS5091, dose 2; Drug2: Placebo Healthy subjects
  Interventions: Drug: HRS5091
- Part 1a Treatment group 3 (Experimental): Intervention: Drug1: HRS5091, dose 3; Drug2: Placebo Healthy subjects
  Interventions: Drug: HRS5091
- Part 1a Treatment group 4 (Experimental): Intervention: Drug1: HRS5091, dose 4; Drug2: Placebo Healthy subjects
  Interventions: Drug: HRS5091
- Part 1a Treatment group 5 (Experimental): Intervention: Drug1: HRS5091, dose 5; Drug2: Placebo Healthy subjects
  Interventions: Drug: HRS5091
- Part 1b Treatment group 3 (Experimental): Intervention: Drug1: HRS5091, dose 3; Drug2: Placebo Healthy subjects Food effect
  Interventions: Drug: HRS5091
- Part 1c Treatment group 6 (Experimental): Intervention: Drug1: HRS5091, dose 3; Drug2: Placebo Healthy subjects
  Interventions: Drug: HRS5091
- Part 2 Treatment group 7 (Experimental): Intervention: Drug1: HRS5091, dose 3; Drug2: Placebo CHB subjects
  Interventions: Drug: HRS5091
- Part 2 Treatment group 8 (Experimental): Intervention: Drug1: HRS5091, dose 4; Drug2: Placebo CHB subjects
  Interventions: Drug: HRS5091
- Part 2 Treatment group 9 (Experimental): Intervention: Drug1: HRS5091, dose 5; Drug2: Placebo CHB subjects
  Interventions: Drug: HRS5091

INTERVENTIONS:
Drug: HRS5091 — Single dose in group 1-5
  Multiple doses in group 6-9
  Other Names: Placebo

SUMMARY:
The study is a randomized, Double-Blind, Placebo-Controlled study to evaluate the safety, tolerability and pharmacokinetics, pharmacodynamics and food effect of HRS5091. The study will be conducted in three parts sequentially:

Part 1a will consist of 58 healthy subjects, 5 groups. The purpose of this part is to explore the safety, tolerability and pharmacokinetics of single doses of HRS5091 tablet in healthy subjects.

Part 1b will consist of 18 healthy subjects and it is one of groups in Part 1a.The purpose of this part is to explore food effect of HRS5091 in healthy subjects.

Part 1c will consist of 10 healthy subjects, 1 groups. The purpose of this part is to explore the safety, tolerability and pharmacokinetics of multiple doses of HRS5091 tablet in healthy subjects.

Part 2 will consist of 30 CHB patients.The purpose of this part is to explore the safety, tolerability and pharmacokinetics, pharmacodynamics of multiple doses of HRS5091 tablet in naïve and treatment-discontinued chronic hepatitis B (CHB) patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

  1. Signed informed consent.
  2. Aged 18~55.
  3. Body weight ≥ 50 kg for male; ≥ 45 kg for female, body mass index (BMI) between 18 to 28 kg/m².
  4. Vital signs, physical examination, laboratory results are within normal range or considered not clinically significant.
  5. Female subjects (including partner) of childbearing potential must be using a medically acceptable form of birth control.
* CHB subjects

  1. Signed informed consent.
  2. Aged 18~65.
  3. CHB subjects should meet one of the following two criteria:

     * IgM(immunoglobulin M) HBcAb negative and HBsAg positive.
     * Two recorded HBsAg positive, and the time interval between the two tests was at least 6 months, one of which was the result of this screening
  4. CHB subjects should also meet the following criteria:

     * No treatment with nucleosides analogues or discontinued treatment with nucleosides analogues least 6 months at screening
     * Have not received interferon therapy or discontinued treatment with interferon analogues least 3 months at screening
     * HBeAg positive，HBV(hepatitis B virus) DNA≥ 20000 IU/mL; HBeAg negative, HBV DNA≥ 2000 IU/mL
     * ALT(Alanine aminotransferase)> 1 ULN(upper limit of normal) by two measurements within 6 months before enrollment.The interval between two measurements shall exceed 14 days;
  5. Female subjects (including partner) of childbearing potential must be using a medically acceptable form of birth control.

Exclusion Criteria:

* Healthy subjects

  1. Currently suffering from cardiovascular, liver, kidney, digestive, nervous, blood, thyroid or mental diseases.
  2. Have a digestive system disease or a medical history of severe digestive system disease at present or in the past month.
  3. Have severe infection, severe trauma or major surgical operations within 3 months. Plan to receive surgery during the trial and within two weeks after the end of the trial.
  4. 12-ECG test have clinical significant abnormality or the QT interval (QTc) > 470 ms(male)/QTc)> 480 ms(male) or<300ms(female).
  5. Have a medical history of immune-mediated diseases.
  6. Screening for infectious diseases is positive,Including HBsAg, Anti-HCV(hepatitis C virus), TPPA(Treponema pallidum particle agglutination assay), Anti-HIV.Treponema pallidum antibody screen positive, at the investigator's discretion in conjunction with RPR(rapid plasma reagin assay) results.
  7. Suspected allergy to any ingredient in the study drug.
  8. Have any drug that inhibits or induces liver metabolism within 1 month.
  9. Take any prescription drugs, over-the-counter drugs and Chinese herbal medicines within 14 days before taking the study drug, or plan to take other drugs during the test period.
  10. Participated in clinical trials of any drug or medical device within 3 months before screening.
  11. Had donated blood/blood transfusion≥ 200 mL within 1 months prior to screening or donated blood or blood transfusion≥ 450 mL within 3 months prior to screening.
  12. The average daily smoking ≥ 5 cigarettes within three months; the average daily alcohol intake in a month exceeds 15 g (15 g alcohol is equivalent to 450 mL beer or 150 mL wine or 50 mL low-alcohol);
  13. Keep smoking, drinking alcohol or consuming caffeinated foods or beverages (more than 8 cups, 1 cup = 250 mL) 2 days before taking the study drug and during the study; and those who have special dietary requirements and cannot follow the unified diet;
  14. Pregnant or lactating women;
  15. Drug screening or alcohol breath test is positive.
  16. Other conditions that the investigator believes the subject is not suitable.
* CHB subjects

  1. Currently suffering from serious cardiovascular, liver, kidney, digestive, nervous, blood, thyroid or mental diseases other than hepatitis B.
  2. People have acute or chronic liver disease by non-HBV infection (Whether fatty liver is excluded or not is determined by the investigator).
  3. Liver stiffness (LSM)> 12.4 kPa(kilopascal) by noninvasive transient liver elastography (eg Fibroscan®) or recorded liver biopsy suggesting cirrhosis or extensive fibrosis within 6 months before randomization.
  4. Primary liver cancer, high-risk groups of primary liver cancer or AFP(alpha fetoprotein)> 50g/L;
  5. Have clinically demonstrated or history of liver function decompensation, including but not limited to: hepatic encephalopathy, hepatorenal syndrome, splenomegaly, ascites, etc.;
  6. Laboratory inspection:

     1. Platelet count <90×10⁹/L;
     2. White blood cell count <3.0×10⁹/L;
     3. Absolute value of neutrophils <1.5×10⁹/L;
     4. Serum total bilirubin>2×ULN;
     5. Albumin <30 g/L;
     6. Creatinine clearance rate ≤60ml/min;
     7. INR(international normalized ratio)>1.5;
     8. ALT> 5 ULN on screening/baseline visit
  7. HIV and/or syphilis antibody positive (Treponema pallidum antibody screen positive, at the investigator's discretion in conjunction with RPR results).
  8. Subjects who have previously received organ/bone marrow transplantation;
  9. Have used immunosuppressants, immunomodulators or cytotoxic drugs within 6 months before the study medication;
  10. Suspected allergy to any ingredient in the study drug.
  11. 12-ECG test have clinical significant abnormality or the QT interval (QTc) > 470 ms(male)/QTc)> 480 ms(male) or<300ms(female).
  12. The average daily smoking ≥ 5 cigarettes within three months; the average daily alcohol intake in a month exceeds 15 g (15 g alcohol is equivalent to 450 mL beer or 150 mL wine or 50 mL low-alcohol);
  13. Keep smoking, drinking alcohol or consuming caffeinated foods or beverages (more than 8 cups, 1 cup = 250 mL) 2 days before taking the study drug and during the study; and those who have special dietary requirements and cannot follow the unified diet;
  14. Pregnant or lactating women;
  15. Drug screening or alcohol breath test is positive.
  16. Other conditions that the investigator believes the subject is not suitable.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-11-23 (Estimated); Study Completion 2021-11-23 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of treatment-related | 29 DAYS for Group 1.2.4.5; 58 DAYS for Group 3; 42 DAYS for Group 6；56 DAYS for Group 7-9；
  adverse events as assessed by CTCAE v5.0
Maximum Plasma Concentration [Cmax] | 0-672 hours after each dose for Group 1-9
  Pharmacokinetic parameters of HRS5091, main metabolite and identified major metabolites in plasma
Area under the concentration time curve [AUC] | 0-672 hours after each dose for Group 1-9
  Pharmacokinetic parameters of HRS5091, main metabolite and identified major metabolites in plasma
Time to maximum plasma concentration [Tmax] | 0-672 hours after each dose for Group 1-9
  Pharmacokinetic parameters of HRS5091, main metabolite and identified major metabolites in plasma
Apparent clearance [CL/F] | 0-672 hours after each dose for Group 1-9
  Pharmacokinetic parameters of HRS5091, main metabolite and identified major metabolites in plasma
Half-time [t1/2] | 0-672 hours after each dose for Group 1-9
  Pharmacokinetic parameters of HRS5091, main metabolite and identified major metabolites in plasma
Apparent volume of distribution [Vz/F(Vd)] | 0-672 hours after each dose for Group 1-9
  Pharmacokinetic parameters of HRS5091, main metabolite and identified major metabolites in plasma
Mean retention time [MRT] | 0-672 hours after each dose for Group 1-9
  Pharmacokinetic parameters of HRS5091, main metabolite and identified major metabolites in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China